CLINICAL TRIAL: NCT01573130
Title: An Internet-administered, Therapist-supported Physical Exercise Program for the Treatment of Depression
Brief Title: Treating Depression With Physical Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Per Carlbring, PhD, Professor, Umeå University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Progredi
Record Dates: First submitted 2012-03-31; First posted 2012-04-06 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Depression
Keywords: Depression; Physical exercise; Internet
MeSH Terms: conditions — Depression; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Initial treatment group (Experimental): Group receives treatment.
  Interventions: Behavioral: Physical exercise program
- Waiting list control group (No Intervention): The waiting list control group receives treatment after 9 weeks, before which they do weekly ratings.

INTERVENTIONS:
Behavioral: Physical exercise program — An individualized physical exercise program, administered per internet. Some therapist-support will also be included.
  Arms: Initial treatment group

SUMMARY:
The purpose of the study is to investigate the effects of an internet-administered, therapist-assisted physical exercise program for the treatment of depression.

DETAILED DESCRIPTION:
Previous research has found promising results regarding physical exercise as treatment of depression. This study will test a 9 week, internet-administered, therapist-assisted physical exercise program.

ELIGIBILITY:
Inclusion Criteria:

* Satisfy DSM-IV criteria for depression
* Living in Sweden and being able to read Swedish
* Access to computer with internet connection

Exclusion Criteria:

* Currently receiving other psychological treatment
* Non-stable use of psychoactive medication
* Deemed to suffer from a too severe depression, or being suicidal
* Deemed to suffer from other psychological disorder, e.g. psychosis, bipolarity etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-06 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) | 24 hours
  9-item depression rating scale.
Change from baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) | 6 months
  9-item depression rating scale.
Change from baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) | Week 1 of treatment duration
  9-item depression rating scale.
Change from baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) | Week 2 of treatment duration
  9-item depression rating scale.
Change from baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) | Week 3 of treatment duration
  9-item depression rating scale.
Change from baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) | Week 4 of treatment duration
  9-item depression rating scale.
Change from baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) | Week 5 of treatment duration
  9-item depression rating scale.
Change from baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) | Week 6 of treatment duration
  9-item depression rating scale.
Change from baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) | Week 7 of treatment duration
  9-item depression rating scale.
Change from baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) | Week 8 of treatment duration
  9-item depression rating scale.

SECONDARY OUTCOMES:
Change from baseline in Beck Depression Inventory (BDI) | 24 hours
  21 item rating scale for depression symptoms.
Change from baseline in Beck Depression Inventory (BDI) | 6 months
  21 item rating scale for depression symptoms.
Change from baseline in Beck Anxiety Inventory (BAI) | 24 hours
  21 item rating scale for anxiety symptoms.
Change from baseline in Beck Anxiety Inventory (BAI) | 6 months
  21 item rating scale for anxiety symptoms.
Change from baseline in Quality Of Life Inventory (QOLI) | 24 hours
  The QOLI assessment yields an overall score and a profile of problems and strengths in 16 areas of life such as love, work and play. The QOLI test is a measure of positive psychology and positive mental health.
Change from baseline in Quality Of Life Inventory (QOLI) | 6 months
  The QOLI assessment yields an overall score and a profile of problems and strengths in 16 areas of life such as love, work and play. The QOLI test is a measure of positive psychology and positive mental health.
Change from baseline in Patient Health Questionnaire (PHQ-9) | 24 hours
  The PHQ-9 is the nine item depression scale of the Patient Health Questionnaire. The PHQ-9 is a powerful tool for assisting primary care clinicians in diagnosing depression as well as selecting and monitoring treatment. The PHQ-9 is based directly on the diagnostic criteria for major depressive disorder in the Diagnostic and Statistical Manual Fourth Edition (DSM-IV).
Change from baseline in Patient Health Questionnaire (PHQ-9) | 6 months
  The PHQ-9 is the nine item depression scale of the Patient Health Questionnaire. The PHQ-9 is a powerful tool for assisting primary care clinicians in diagnosing depression as well as selecting and monitoring treatment. The PHQ-9 is based directly on the diagnostic criteria for major depressive disorder in the Diagnostic and Statistical Manual Fourth Edition (DSM-IV).
Change from baseline in the International Physical Activity Questionnaire (IPAQ) | 24 hours
  The International Physical Activity Questionnaire is a measure of physical activity.
Change from baseline in the International Physical Activity Questionnaire (IPAQ) | 6 months
  The International Physical Activity Questionnaire is a measure of physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Per Carlbring, Professor, Principal Investigator — Department of Psychology, Umeå University
Locations (1):
- Department of Psychology, Umeå University, Umeå, Västerbotten County, Sweden

REFERENCES:
- [Result] Strom M, Uckelstam CJ, Andersson G, Hassmen P, Umefjord G, Carlbring P. Internet-delivered therapist-guided physical activity for mild to moderate depression: a randomized controlled trial. PeerJ. 2013 Oct 3;1:e178. doi: 10.7717/peerj.178. eCollection 2013. PMID 24109561